CLINICAL TRIAL: NCT01210248
Title: Correlation Between CYP2C19 Genotype, Level Of Clopidogrel Metabolite And Platelet Inhibition Status
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: NO 51/10
Record Dates: First submitted 2010-09-26; First posted 2010-09-28 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-05

CONDITIONS: PRIMARY FOCUS:PATIENT THAT TAKE CLOPIDOGREL
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: BLOOD COLLECTION — BLOOD SAMPLE WILL BE COLLECTED FOR 3 KINDS OF TESTS

SUMMARY:
The aim of this study is to check correlation between CYP2C19 genotype level of clopidogrel metabolite in plasma and platelet inhibition status.

DETAILED DESCRIPTION:
THE FIRST PHASE OF THE RESEARCH WILL INVOLVE PATIENTS RECRUITMENT AND INFORMED CONSENT FOR GENETIC TESTING.THE MAJORITY OF PATIENTS WILL BE RECRUITED FROM EMERGENCY DEPARTMENT. EVERY PATIENT WILL BE ASKED ABOUT HIS AND HIS PARENT'S ETHNICITY (ASHKENASI OR SEPHARDY JEW) AND ADDITIONAL DRUGS HE TAKES. IF PATIENT AGREES TO PARTICIPATE IN THE STUDY , HIS BLOOD SAMPLE WILL BE COLLECTED FOR 3 KINDS OF TESTS:

1. GENETIC (FOR CYP450 2C19)
2. PLATELET MAPPING TEST ( BY THROMBOELASTOGRAPH ASSAY)
3. CLOPIDOGREL INACTIVE METABOLITE DETERMINATION BY CHROMATOGRAPHIC METHOD

ELIGIBILITY:
Inclusion Criteria:

* > 18 OLD PATIENTS
* THAT TAKE CLOPIDOGREL MORE THAN 1 WEEK

Exclusion Criteria:

* PREGNANCY
* CHRONIC LIVER DISEASES

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: THE RESEARCH WILL INVOLVE PATIENTS THAT TAKE CLOPIDOGREL AND READY TO GIVE INFORMED CONSENT FOR GENETIC TESTING.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-01

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center, Zeriffin, Israel, Israel